CLINICAL TRIAL: NCT02535182
Title: Pilot Study Using Propranolol To Promote Prenylation Of The Gtpase Rap1b In Hematopoietic Stem Cell Transplant Recipients
Brief Title: Pilot Study Using Propranolol To Promote Prenylation Of Gtpase Rap1b In Hematopoietic Stem Cell Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jennifer M. Knight, Assistant Professor, Medical College of Wisconsin
Other Study IDs: 24391
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMCs) will be isolated from the whole blood samples collected from patients at the three designated time points (Baseline, Day -2, and Day +28). Members of Dr. Carol Williams' laboratory (Professor, Pharmacology and Toxicology, MCW) will conduct western blotting on the cytosolic and membrane fractions of isolated PBMCs to determine the distribution of Rap1 in the different fractions, and the status of Rap1 prenylation in the cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Arm: Patients who participate as controls on the main study will be controls on this ancillary study. The control arm will have blood drawn at baseline, day -2 and day -28 for the Rap1 testing.
  Interventions: Other: Blood Draw
- Propranolol Arm: Patients who participate on the propranolol arm on the main study will be on the propranolol arm on this ancillary study. The propranolol arm will have blood drawn at baseline, day -2 and day -28 for the Rap1 testing.
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Lab will draw one tube of blood to be stored in 8 mL Becton Dickinson (BD) Vacutainer Cell Preparation Tube (CPT) tubes at three study time points as described in Table 4.7b. These time points include baseline, Day -2 (immediately prior to transplant, central line placement, or administration of any conditioning regimen), and Day +28.
  Peripheral blood mononuclear cells (PBMCs) will be isolated from the whole blood samples collected from patients at the three designated time points (Baseline, Day -2, and Day +28). The lab will conduct western blotting on the cytosolic and membrane fractions of isolated PBMCs to determine the distribution of Rap1 in the different fractions, and the status of Rap1 prenylation in the cells.

SUMMARY:
This is a an ancillary study designed to explore whether an additional cell signaling pathway (prenylation of Rap1) that was recently identified as being under beta-adrenergic control may be affected by beta-blocker use.

DETAILED DESCRIPTION:
This is a proof of concept randomized controlled pilot study assessing whether prenylation and membrane localization of Rap1 in PBMCs can be altered in individuals undergoing autologous Hematopoietic Cell Transplant (HCT) for Multiple Myeloma by administering a daily beta-blocker (propranolol) to 20 participants. Outcomes of patients on this clinical trial will be compared to 20 participants in a control arm.

ELIGIBILITY:
Inclusion Criteria:

Patients with multiple myeloma receiving an autologous HCT are eligible when the following criteria are met:

1. 18-75 years of age
2. ≤ 1 year since initiation of systemic anti-myeloma therapy
3. Patient is scheduled for autologous hematopoietic stem cell transplant as the upfront therapy for their multiple myeloma
4. Karnofsky Performance Status of ≥90 %; patients eligible for HCT are eligible for the study
5. All men and women must agree to practice effective contraception during the study period if not otherwise documented to be infertile.

Exclusion Criteria:

1. Prior autologous HCT
2. Non secretory multiple myeloma
3. Concurrent beta-blocker therapy at or within 3 weeks of study entry.
4. Previous intolerance to beta-blocker therapy
5. Any medical contraindications to beta-blocker therapy including, but not limited to, symptomatic hypotension; drug hypersensitivity; sinus bradycardia, sick sinus syndrome, or 2nd or 3rd degree atrioventricular block without a pacemaker; uncompensated heart failure; or uncontrolled asthma
6. Active, untreated depression screened for by the HCT physician (Patients who screen positive will be offered a referral to the MCW Psycho-Oncology program for further evaluation and treatment)
7. Concurrent use of medications as specified in the protocol throughout the study or within one week of study entry.
8. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are enrolled in the parent study (NCT02420223) are eligible for this ancillary study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Prenylation levels in response to propranolol in a population of patients undergoing autologous hematopoietic stem cell transplantation | 1 year
  Level of prenylation will be compared between patients exposed vs. not exposed to propranolol from 1-3 weeks before to 4 weeks following transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knight, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT02535182/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT02535182/ICF_001.pdf